CLINICAL TRIAL: NCT03692221
Title: Percutaneous Image Guided Delivery of Autologous Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Symptomatic Degenerated Intervertebral Disc Disease
Brief Title: Mesenchymal Stem Cells for Lumbar Degenerative Disc Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Stalled due to Covid
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Salim M Hayek, MD, PhD, Chief, Division of Pain Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 014924/0012/A002
Record Dates: First submitted 2018-09-24; First posted 2018-10-02 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Disc Degeneration
Keywords: Back pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Intervention Model Description: 24 participants will be equally randomized into two groups; 12 Healthy controls subjects & 12 treatment subjects. The treatment group will then be sub-divided and randomized into 6 subjects receiving a low dosage treatment and 6 subjects receiving a high dosage treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MSC treatment group 1 (Experimental): Low dose of Autologous Bone Marrow Derived Mesenchymal Stem Cells (MSC) -A one time injection of 1-2 ml of 2 x 106/ml concentrated solution
  Interventions: Drug: MSC Treatment group 1 (low dose)
- MSC treatment group 2 (Active Comparator): High dose of Autologous Bone Marrow Derived Mesenchymal Stem Cells (MSC) -A one time injection of 1-2 ml of 4 x 106/ml concentrated solution
  Interventions: Drug: MSC Treatment group 2 (high dose)
- Healthy Control (no treatment) (Active Comparator): Comparative analysis of psychometric and morphometric based data
  Interventions: Other: Healthy Control (no treatment)

INTERVENTIONS:
Drug: MSC Treatment group 1 (low dose) — Autologous Bone Marrow Derived Mesenchymal Stem Cells (MSC) - A one time injection of 1-2 ml of a 4 x 106/ml concentration solution
  Arms: MSC treatment group 1
Drug: MSC Treatment group 2 (high dose) — Autologous Bone Marrow Derived Mesenchymal Stem Cells (MSC) - A one time injection of 1-2 ml of a 4 x 106/ml concentration solution
  Arms: MSC treatment group 2
Other: Healthy Control (no treatment) — Comparative analysis of psychometric and morphometric based data
  Arms: Healthy Control (no treatment)

SUMMARY:
This study seeks to bridge these technologies and obtain data regarding the safety and efficacy of image guided percutaneous needle injection of expanded autologous bone marrow derived mesenchymal stem cells to symptomatic degenerated intervertebral discs in humans. The primary outcome will be to assess the safety and efficacy and monitor for adverse events.

DETAILED DESCRIPTION:
Bone Marrow Aspiration and Cell Culture Procedure

Utilizing fluoroscopic guidance, a coaxial needle will be advanced to the bone marrow space. The inner portion will be removed and 10-20mL of marrow aspirated.

MSCs will be isolated and cultured in the Case Western Reserve University National Center for Regenerative Medicine/Seidman Cancer Center Cellular Therapy Lab using standard operating procedures established under the ongoing IND - as above.

MSC Delivery/Transplantation Procedure

Utilizing fluoroscopic guidance, a needle will be advanced to the outer annulus of the affected disc(s). Through the coaxial anchor, a needle will be advanced to the middle 1/3 of the disc, and confirmed in two planes (AP and lateral).

On the day of infusion, MSCs will be transported from the Cellular Therapy Lab to the IR suite in a validated dry shipper. MSCs will be thawed in a 37ºC water bath and drawn into 1 ml syringes. Prior to delivery, an aliquot of the infused product will be tested for viability (trypan blue exclusion). Viability must be >70% for cell transplantation. Treatment group one will receive an injection of 1-2 ml of a 2 x 106/ml concentration solution of MSCs and treatment group 2 will 1-2 ml of a 4 x 106/ml concentration solution of MSCs. Both treatment groups will be injected under intermittent fluoroscopic observation. A manometer will be used to monitor disc pressures, especially during MSC injection keeping pressure below 100 psi. Specifically, the volume of injectate will be determined based on three dynamic factors: real time imaging of contained contrast volume during discography, psi as measured during the injection (< 100), and patient's symptoms (if patient's pain exceeds baseline, injection will be stopped) - up to a volume of 2cc of the assigned concentration.

An aliquot of infused product will be submitted to the University Hospitals Cleveland Medical Center Microbiology Laboratory to test for microbiological contamination. In the event of a positive microbial test following administration of a cellular product: 1) The Principal Investigator and his/her designee will be notified and will notify the participant, 2) The contaminant will identified to a species level and antibiotic sensitivities determined, 3) The Medical Director of the Cellular Therapy Laboratory and/or the Principal Investigator will determine the best course of action based on the clinical situation. This may include blood cultures, administration of prophylactic antibiotics, and repeat cultures on the cell product. 4) An investigation to determine the source of the contamination will be conducted, and appropriate corrective measures will be undertaken. Finally, the adverse event will be reported to the IRB and FDA based on the respective federal and institutional reporting requirement, as well the approved data safety monitoring board charter.

MRI/Quantitative MRI Procedure

Routine images of the lumbar spine (sagittal and axial T1 and T2 weighted images) will be obtained for the purposes of: Monitoring for potential alternative effects of the cells including osteophyte formation, as well as any unexpected local outcome. In addition, a quantative MRI including fingerprinting. Magnetic resonance Fingerprinting (MRF) allows rapid and simultaneous quantification of T1and T2 relaxation times. The MRF sequence is based on varying multiple MR acquisition parameters [ e.g. flip angle (FA) and time of repetition (TR)] in a pseudorandom manner, such that unique signal evolutions called "fingerprints" are generated for each combination of tissue properties. These fingerprints are compared with a dictionary of simulated fingerprints generated for that sequence by a pattern matching process. Once there is a pattern match, the T1 and T2 values used to generate that dictionary entry are assigned to that voxel and used to create T1 and T2 maps that are perfectly anatomically co-registered.

For spine, the proposed MRF sequence is based on a multislice Fast Imaging with Steady Precession (FISP) acquisition. Scanning will be done both in sagittal and axial planes using a multislice acquisition. The scan parameters are as follows:

FOV: 400 mm, matrix 400 x 400 mm , TR/TE: 13-15 msec, in-plane resolution 1 x 1 mm, section thickness 5 mm, flip angle 5-75 degrees, acquisition time ~ 39 seconds per slice, with ~ 4 minutes scan time for a 5 slice sagittal image. In axial plane, the disc would be covered at each intervertebral level in 4-5 transverse slices and each axial acquisition would take ~ 3 minutes scan time.

The MRF maps would be directly generated as DICOM images using Gadgetron online reconstruction. Image analysis would be done using a DICOM viewing software to draw Regions of Interest (ROIs) on nucleus pulposus for direct quantification of relaxation times. There is the capacity to generate MRF maps from raw data on Matlab which can also be used to draw ROIs for simultaneous quantification of T1 and T2 relaxation times.

These values will be calculated on the pre and post treatment MRIs.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms despite conservative (non-surgical) management for > 6 months

  * Leg pain, if present, is of nonradicular origin, i.e., not due to stimulation of nerve roots or dorsal root ganglion of a spinal nerve by compressive forces.
  * Leg pain, if present, does not extend below the knee and is no greater than 50% of low back pain as measured on a visual analog scale. If bilateral leg pain existed, the worst leg pain is no greater than 50% of low back pain.
* Diagnostic medical branch block or facet joint injection between 18 months and 2 weeks prior to the study procedure indicates no facet joint involvement.
* Distress and risk assessment method stratification to a) normal or b) at risk designations
* Modified Pfirrmann MR classification of implicated intervertebral discs of III, IV, or V
* Absence of infection
* Absence of coagulopathy
* Ability to provide informed written consent

Exclusion Criteria:

* Age > 80y or < 18 y
* Neoplasia
* History of recent or active malignancy(non-melanoma skin cancers, carcinoma in situ, etc. are allowable)
* Active infection
* Underlying congenital segmentation or other spinal anomalies that result in differential intervertebral disc pressures
* Significant spinal stenosis

  * Interpreted as "severe" on any cross sectional imaging study
* Pregnant or planning to become pregnant
* Contraindication to MRI

  * Indwelling medical devices such as pacemakers, aneurysm clips, etc
  * Indwelling metal from any other cause (trauma, etc)

    * To be excluded with history and radiographs, as necessary
* Immunosuppression
* History or laboratory results indicative of any significant cardiac, endocrine, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neoplastic, or other disorder that in the opinion of the Principal Investigator or his/her designee would preclude the safe performance of BM aspiration, transplantation of autologous MSCs, or performance of any of the planned study assessments.
* Uncorrectable coagulopathies
* Concurrent participation in another investigational trial involving systemic administration of agents or within the previous 30 days.
* Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI >35).
* Clinically relevant instability on flexion-extension as determined by the investigator by overlaying films.
* Have undergone a previous surgery at the involved level that may have altered the target disc (e.g. discectomy, laminectomy, foraminotomy, fusion, intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation etc.).
* Have an acute fracture of the spine at the time of enrollment in the study. Clinically compromised vertebral bodies at the affected level due to current or past trauma, e.g., sustained pathological fracture or multiple fractures of vertebrae.
* Have a history of epidural steroid injections within 1 week prior to study treatment.
* Have received chronic (more than 7 consecutive days) treatment with systemic corticosteroids at a dose equivalent to prednisone ≥ 10 mg/day within 14 days prior to injection procedure.
* Have received systemic or local nonsteroidal anti-inflammatory drugs (NSAIDS) injections into the index and/or adjacent vertebral levels within 48 hours prior to study procedure.
* Have a known history of hypersensitivity or anaphylactic reaction to murine or bovine products or dimethyl sulfoxide (DMSO).
* Have a known history of hypersensitivity or anaphylactic reaction to products from birds, such as feathers, eggs or poultry.
* Have a positive screen for human immunodeficiency virus (HIV) by antibodies or nucleic acid test.
* Have had treatment with any investigational therapy or device within 6 months of study procedure and/or plans to participate in any other allogeneic stem cell/progenitor cell therapy trial during the 3-year follow-up period.
* Have been a recipient of prior stem cell/progenitor cell therapy or other biological intervention to repair the target intervertebral disc.
* Are transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program.
* Habitual use of tobacco throughout the trial and follow-up.
* Have a mental illness that could prevent completion of the study or protocol questionnaires. If subjects with psychiatric disease are stable, then they should be allowed to participate in the trial.
* Neurological diseases including unstable diseases or disease which renders subjects unable to give informed consent which renders unable to give informed consent. (Subjects with well controlled epilepsy should not be excluded.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment related adverse events | From baseline/randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
  assessing for worsening of patients' baseline symptoms or functions (will be considered an AE); (also general AE events), particularly AE events related to the procedures/treatment. All AEs will be assessed by common terminology criteria for adverse events. .

SECONDARY OUTCOMES:
Changes in Pain -Visual Analogue Scale (VAS) for back pain | Baseline, 1 month, 6 months and 1 year
  Temporal evaluation of pain before and after the procedure will be analyzed through documentation of Visual Analogue Scale of back pain (VAS).
  The VAS is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is a unidimensional measure of pain intensity The instrument is presented by a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. No pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) (11).
Changes in Pain - Oswestry Disability Index (ODI) scores over time | Baseline, 1 month, 6 months and 1 year
  Temporal evaluation of pain before and after the procedure will be analyzed through documentation of Oswestry Disability Index (ODI) scores over time. Scoring - For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated. Interpretation scores go from minimal 0% disability to 100% disability.
changes in Quality of life - Short form Health Survey 36 (SF-36) | Baseline, 1 month, 6 months and 1 year
  Temporal evaluation of quality of life before and after the procedure will be analyzed through documentation of SF36 quality of life questionnaire scores. Although this study is not cancer related, this questionnaire is a validated instrument for the evaluation of treatment related impact on quality of life - a critical outcome measure. Scoring - consisting of eight scaled scores which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
changes in MRI monitoring of transplant site | Baseline and 1 year, if a subject were to withdraw prior to completion of the study and received MSC an MRI with be obtained.
  Magnetic resonance T2 mapping will be performed on all discs undergoing treatment for evaluation of potential quantitative, reproducible imaging change following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Lawrence, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker J 3rd, El Abd O, Isaac Z, Muzin S. Discography in practice: a clinical and historical review. Curr Rev Musculoskelet Med. 2008 Jun;1(2):69-83. doi: 10.1007/s12178-007-9009-9. PMID 19468876
- [Background] Frymoyer JW, Cats-Baril WL. An overview of the incidences and costs of low back pain. Orthop Clin North Am. 1991 Apr;22(2):263-71. PMID 1826550
- [Background] Cheung KM, Karppinen J, Chan D, Ho DW, Song YQ, Sham P, Cheah KS, Leong JC, Luk KD. Prevalence and pattern of lumbar magnetic resonance imaging changes in a population study of one thousand forty-three individuals. Spine (Phila Pa 1976). 2009 Apr 20;34(9):934-40. doi: 10.1097/BRS.0b013e3181a01b3f. PMID 19532001
- [Background] Madigan L, Vaccaro AR, Spector LR, Milam RA. Management of symptomatic lumbar degenerative disk disease. J Am Acad Orthop Surg. 2009 Feb;17(2):102-11. doi: 10.5435/00124635-200902000-00006. PMID 19202123
- [Background] Bogduk N, Karasek M. Two-year follow-up of a controlled trial of intradiscal electrothermal anuloplasty for chronic low back pain resulting from internal disc disruption. Spine J. 2002 Sep-Oct;2(5):343-50. doi: 10.1016/s1529-9430(02)00409-6. PMID 14589465
- [Background] Kvarstein G, Mawe L, Indahl A, Hol PK, Tennoe B, Digernes R, Stubhaug A, Tonnessen TI, Beivik H. A randomized double-blind controlled trial of intra-annular radiofrequency thermal disc therapy--a 12-month follow-up. Pain. 2009 Oct;145(3):279-286. doi: 10.1016/j.pain.2009.05.001. Epub 2009 Aug 3. PMID 19647940
- [Background] Freeman BJ, Fraser RD, Cain CM, Hall DJ, Chapple DC. A randomized, double-blind, controlled trial: intradiscal electrothermal therapy versus placebo for the treatment of chronic discogenic low back pain. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2369-77; discussion 2378. doi: 10.1097/01.brs.0000186587.43373.f2. PMID 16261111
- [Background] Williams JD, P.K., ed. Lower Back Pain and Disorders of Intervertebral Discs. 11 ed. Campbell's Operative Orthopaedics., ed. C.a. Beaty. 2007, Mosby.
- [Background] Hilibrand AS, Robbins M. Adjacent segment degeneration and adjacent segment disease: the consequences of spinal fusion? Spine J. 2004 Nov-Dec;4(6 Suppl):190S-194S. doi: 10.1016/j.spinee.2004.07.007. PMID 15541666
- [Background] Nesti LJ, Li WJ, Shanti RM, Jiang YJ, Jackson W, Freedman BA, Kuklo TR, Giuliani JR, Tuan RS. Intervertebral disc tissue engineering using a novel hyaluronic acid-nanofibrous scaffold (HANFS) amalgam. Tissue Eng Part A. 2008 Sep;14(9):1527-37. doi: 10.1089/ten.tea.2008.0215. PMID 18707229
- [Background] Shuff C, An HS. Artificial disc replacement: the new solution for discogenic low back pain? Am J Orthop (Belle Mead NJ). 2005 Jan;34(1):8-12. PMID 15707133
- [Background] Solchaga LA, Penick K, Goldberg VM, Caplan AI, Welter JF. Fibroblast growth factor-2 enhances proliferation and delays loss of chondrogenic potential in human adult bone-marrow-derived mesenchymal stem cells. Tissue Eng Part A. 2010 Mar;16(3):1009-19. doi: 10.1089/ten.TEA.2009.0100. PMID 19842915
- [Background] Wang F, Dennis JE, Awadallah A, Solchaga LA, Molter J, Kuang Y, Salem N, Lin Y, Tian H, Kolthammer JA, Kim Y, Love ZB, Gerson SL, Lee Z. Transcriptional profiling of human mesenchymal stem cells transduced with reporter genes for imaging. Physiol Genomics. 2009 Mar 3;37(1):23-34. doi: 10.1152/physiolgenomics.00300.2007. Epub 2008 Dec 30. PMID 19116247
- [Background] Love Z, Wang F, Dennis J, Awadallah A, Salem N, Lin Y, Weisenberger A, Majewski S, Gerson S, Lee Z. Imaging of mesenchymal stem cell transplant by bioluminescence and PET. J Nucl Med. 2007 Dec;48(12):2011-20. doi: 10.2967/jnumed.107.043166. Epub 2007 Nov 15. PMID 18006616
- [Background] Welter JF, Solchaga LA, Penick KJ. Simplification of aggregate culture of human mesenchymal stem cells as a chondrogenic screening assay. Biotechniques. 2007 Jun;42(6):732, 734-7. doi: 10.2144/000112451. PMID 17612296
- [Background] Solchaga LA, Temenoff JS, Gao J, Mikos AG, Caplan AI, Goldberg VM. Repair of osteochondral defects with hyaluronan- and polyester-based scaffolds. Osteoarthritis Cartilage. 2005 Apr;13(4):297-309. doi: 10.1016/j.joca.2004.12.016. PMID 15780643
- [Background] Welter JF, Solchaga LA, Stewart MC. High-efficiency nonviral transfection of primary chondrocytes. Methods Mol Med. 2004;100:129-46. doi: 10.1385/1-59259-810-2:129. PMID 15280593
- [Background] Solchaga LA, Welter JF, Lennon DP, Caplan AI. Generation of pluripotent stem cells and their differentiation to the chondrocytic phenotype. Methods Mol Med. 2004;100:53-68. doi: 10.1385/1-59259-810-2:053. PMID 15280587
- [Background] Solchaga LA, Goldberg VM, Caplan AI. Cartilage regeneration using principles of tissue engineering. Clin Orthop Relat Res. 2001 Oct;(391 Suppl):S161-70. doi: 10.1097/00003086-200110001-00016. PMID 11603701
- [Background] Yoo JU, Barthel TS, Nishimura K, Solchaga L, Caplan AI, Goldberg VM, Johnstone B. The chondrogenic potential of human bone-marrow-derived mesenchymal progenitor cells. J Bone Joint Surg Am. 1998 Dec;80(12):1745-57. doi: 10.2106/00004623-199812000-00004. PMID 9875932
- [Background] Lee Z, Dennis JE, Gerson SL. Imaging stem cell implant for cellular-based therapies. Exp Biol Med (Maywood). 2008 Aug;233(8):930-40. doi: 10.3181/0709-MR-234. Epub 2008 May 14. PMID 18480418
- [Background] Richardson SM, Hoyland JA, Mobasheri R, Csaki C, Shakibaei M, Mobasheri A. Mesenchymal stem cells in regenerative medicine: opportunities and challenges for articular cartilage and intervertebral disc tissue engineering. J Cell Physiol. 2010 Jan;222(1):23-32. doi: 10.1002/jcp.21915. PMID 19725073
- [Background] Sobajima S, Vadala G, Shimer A, Kim JS, Gilbertson LG, Kang JD. Feasibility of a stem cell therapy for intervertebral disc degeneration. Spine J. 2008 Nov-Dec;8(6):888-96. doi: 10.1016/j.spinee.2007.09.011. Epub 2007 Dec 21. PMID 18082460
- [Background] Henriksson HB, Svanvik T, Jonsson M, Hagman M, Horn M, Lindahl A, Brisby H. Transplantation of human mesenchymal stems cells into intervertebral discs in a xenogeneic porcine model. Spine (Phila Pa 1976). 2009 Jan 15;34(2):141-8. doi: 10.1097/BRS.0b013e31818f8c20. PMID 19112334
- [Background] Mobasheri A, Csaki C, Clutterbuck AL, Rahmanzadeh M, Shakibaei M. Mesenchymal stem cells in connective tissue engineering and regenerative medicine: applications in cartilage repair and osteoarthritis therapy. Histol Histopathol. 2009 Mar;24(3):347-66. doi: 10.14670/HH-24.347. PMID 19130405
- [Background] Centeno CJ, Busse D, Kisiday J, Keohan C, Freeman M, Karli D. Increased knee cartilage volume in degenerative joint disease using percutaneously implanted, autologous mesenchymal stem cells. Pain Physician. 2008 May-Jun;11(3):343-53. PMID 18523506
- [Background] Sakai D, Mochida J, Iwashina T, Watanabe T, Nakai T, Ando K, Hotta T. Differentiation of mesenchymal stem cells transplanted to a rabbit degenerative disc model: potential and limitations for stem cell therapy in disc regeneration. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2379-87. doi: 10.1097/01.brs.0000184365.28481.e3. PMID 16261113
- [Background] Sakai D, Mochida J, Yamamoto Y, Nomura T, Okuma M, Nishimura K, Nakai T, Ando K, Hotta T. Transplantation of mesenchymal stem cells embedded in Atelocollagen gel to the intervertebral disc: a potential therapeutic model for disc degeneration. Biomaterials. 2003 Sep;24(20):3531-41. doi: 10.1016/s0142-9612(03)00222-9. PMID 12809782
- [Background] Crevensten G, Walsh AJ, Ananthakrishnan D, Page P, Wahba GM, Lotz JC, Berven S. Intervertebral disc cell therapy for regeneration: mesenchymal stem cell implantation in rat intervertebral discs. Ann Biomed Eng. 2004 Mar;32(3):430-4. doi: 10.1023/b:abme.0000017545.84833.7c. PMID 15095817
- [Background] Zhang YG, Guo X, Xu P, Kang LL, Li J. Bone mesenchymal stem cells transplanted into rabbit intervertebral discs can increase proteoglycans. Clin Orthop Relat Res. 2005 Jan;(430):219-26. doi: 10.1097/01.blo.0000146534.31120.cf. PMID 15662327
- [Background] Bendtsen M, Bunger CE, Zou X, Foldager C, Jorgensen HS. Autologous stem cell therapy maintains vertebral blood flow and contrast diffusion through the endplate in experimental intervertebral disc degeneration. Spine (Phila Pa 1976). 2011 Mar 15;36(6):E373-9. doi: 10.1097/BRS.0b013e3181dce34c. PMID 21372649
- [Background] Serigano K, Sakai D, Hiyama A, Tamura F, Tanaka M, Mochida J. Effect of cell number on mesenchymal stem cell transplantation in a canine disc degeneration model. J Orthop Res. 2010 Oct;28(10):1267-75. doi: 10.1002/jor.21147. PMID 20839317
- [Background] See EY, Toh SL, Goh JC. Simulated intervertebral disc-like assembly using bone marrow-derived mesenchymal stem cell sheets and silk scaffolds for annulus fibrosus regeneration. J Tissue Eng Regen Med. 2012 Jul;6(7):528-35. doi: 10.1002/term.457. Epub 2011 Jul 29. PMID 21800436
- [Background] Luo W, Xiong W, Qiu M, Lv Y, Li Y, Li F. Differentiation of mesenchymal stem cells towards a nucleus pulposus-like phenotype utilizing simulated microgravity In vitro. J Huazhong Univ Sci Technolog Med Sci. 2011 Apr;31(2):199. doi: 10.1007/s11596-011-0252-3. Epub 2011 Apr 20. PMID 21505985
- [Background] Yang H, Wu J, Liu J, Ebraheim M, Castillo S, Liu X, Tang T, Ebraheim NA. Transplanted mesenchymal stem cells with pure fibrinous gelatin-transforming growth factor-beta1 decrease rabbit intervertebral disc degeneration. Spine J. 2010 Sep;10(9):802-10. doi: 10.1016/j.spinee.2010.06.019. Epub 2010 Jul 24. PMID 20655810
- [Background] Orozco L, Soler R, Morera C, Alberca M, Sanchez A, Garcia-Sancho J. Intervertebral disc repair by autologous mesenchymal bone marrow cells: a pilot study. Transplantation. 2011 Oct 15;92(7):822-8. doi: 10.1097/TP.0b013e3182298a15. PMID 21792091
- [Background] Yoshikawa T, Ueda Y, Miyazaki K, Koizumi M, Takakura Y. Disc regeneration therapy using marrow mesenchymal cell transplantation: a report of two case studies. Spine (Phila Pa 1976). 2010 May 15;35(11):E475-80. doi: 10.1097/BRS.0b013e3181cd2cf4. PMID 20421856
- [Background] Lazarus HM, Haynesworth SE, Gerson SL, Rosenthal NS, Caplan AI. Ex vivo expansion and subsequent infusion of human bone marrow-derived stromal progenitor cells (mesenchymal progenitor cells): implications for therapeutic use. Bone Marrow Transplant. 1995 Oct;16(4):557-64. PMID 8528172
- [Background] Koc ON, Peters C, Aubourg P, Raghavan S, Dyhouse S, DeGasperi R, Kolodny EH, Yoseph YB, Gerson SL, Lazarus HM, Caplan AI, Watkins PA, Krivit W. Bone marrow-derived mesenchymal stem cells remain host-derived despite successful hematopoietic engraftment after allogeneic transplantation in patients with lysosomal and peroxisomal storage diseases. Exp Hematol. 1999 Nov;27(11):1675-81. doi: 10.1016/s0301-472x(99)00101-0. PMID 10560915
- [Background] Koc ON, Gerson SL, Cooper BW, Dyhouse SM, Haynesworth SE, Caplan AI, Lazarus HM. Rapid hematopoietic recovery after coinfusion of autologous-blood stem cells and culture-expanded marrow mesenchymal stem cells in advanced breast cancer patients receiving high-dose chemotherapy. J Clin Oncol. 2000 Jan;18(2):307-16. doi: 10.1200/JCO.2000.18.2.307. PMID 10637244
- [Background] Koc ON, Lazarus HM. Mesenchymal stem cells: heading into the clinic. Bone Marrow Transplant. 2001 Feb;27(3):235-9. doi: 10.1038/sj.bmt.1702791. PMID 11277170
- [Background] Koc ON, Day J, Nieder M, Gerson SL, Lazarus HM, Krivit W. Allogeneic mesenchymal stem cell infusion for treatment of metachromatic leukodystrophy (MLD) and Hurler syndrome (MPS-IH). Bone Marrow Transplant. 2002 Aug;30(4):215-22. doi: 10.1038/sj.bmt.1703650. PMID 12203137
- [Background] Fibbe WE, Noort WA. Mesenchymal stem cells and hematopoietic stem cell transplantation. Ann N Y Acad Sci. 2003 May;996:235-44. doi: 10.1111/j.1749-6632.2003.tb03252.x. PMID 12799302
- [Background] Lazarus HM, Koc ON, Devine SM, Curtin P, Maziarz RT, Holland HK, Shpall EJ, McCarthy P, Atkinson K, Cooper BW, Gerson SL, Laughlin MJ, Loberiza FR Jr, Moseley AB, Bacigalupo A. Cotransplantation of HLA-identical sibling culture-expanded mesenchymal stem cells and hematopoietic stem cells in hematologic malignancy patients. Biol Blood Marrow Transplant. 2005 May;11(5):389-98. doi: 10.1016/j.bbmt.2005.02.001. PMID 15846293
- [Background] Vadala G, Sowa G, Hubert M, Gilbertson LG, Denaro V, Kang JD. Mesenchymal stem cells injection in degenerated intervertebral disc: cell leakage may induce osteophyte formation. J Tissue Eng Regen Med. 2012 May;6(5):348-55. doi: 10.1002/term.433. Epub 2011 Jun 13. PMID 21671407
- [Background] Foster NE, Thomas E, Bishop A, Dunn KM, Main CJ. Distinctiveness of psychological obstacles to recovery in low back pain patients in primary care. Pain. 2010 Mar;148(3):398-406. doi: 10.1016/j.pain.2009.11.002. Epub 2009 Dec 22. PMID 20022697
- [Background] Maniadakis N, Gray A. The economic burden of back pain in the UK. Pain. 2000 Jan;84(1):95-103. doi: 10.1016/S0304-3959(99)00187-6. PMID 10601677
- [Background] Sakai D. Future perspectives of cell-based therapy for intervertebral disc disease. Eur Spine J. 2008 Dec;17 Suppl 4(Suppl 4):452-8. doi: 10.1007/s00586-008-0743-5. Epub 2008 Nov 13. PMID 19005704
- [Background] Takahashi K, Aoki Y, Ohtori S. Resolving discogenic pain. Eur Spine J. 2008 Dec;17 Suppl 4(Suppl 4):428-31. doi: 10.1007/s00586-008-0752-4. Epub 2008 Nov 13. PMID 19005695
- [Background] Mwale F, Iatridis JC, Antoniou J. Quantitative MRI as a diagnostic tool of intervertebral disc matrix composition and integrity. Eur Spine J. 2008 Dec;17 Suppl 4(Suppl 4):432-40. doi: 10.1007/s00586-008-0744-4. Epub 2008 Nov 13. PMID 19005703
- [Background] Freimark D, Czermak P. Cell-based regeneration of intervertebral disc defects: review and concepts. Int J Artif Organs. 2009 Apr;32(4):197-203. doi: 10.1177/039139880903200403. PMID 19569027
- [Background] Hiyama A, Mochida J, Sakai D. Stem cell applications in intervertebral disc repair. Cell Mol Biol (Noisy-le-grand). 2008 Oct 26;54(1):24-32. PMID 18954548
- [Background] Leung VY, Chan D, Cheung KM. Regeneration of intervertebral disc by mesenchymal stem cells: potentials, limitations, and future direction. Eur Spine J. 2006 Aug;15 Suppl 3(Suppl 3):S406-13. doi: 10.1007/s00586-006-0183-z. Epub 2006 Jul 15. PMID 16845553
- [Background] Cousins JP, Haughton VM. Magnetic resonance imaging of the spine. J Am Acad Orthop Surg. 2009 Jan;17(1):22-30. doi: 10.5435/00124635-200901000-00004. PMID 19136424
- [Background] Kjaer P, Leboeuf-Yde C, Korsholm L, Sorensen JS, Bendix T. Magnetic resonance imaging and low back pain in adults: a diagnostic imaging study of 40-year-old men and women. Spine (Phila Pa 1976). 2005 May 15;30(10):1173-80. doi: 10.1097/01.brs.0000162396.97739.76. PMID 15897832
- [Background] Modic MT, Masaryk TJ, Ross JS, Carter JR. Imaging of degenerative disk disease. Radiology. 1988 Jul;168(1):177-86. doi: 10.1148/radiology.168.1.3289089. No abstract available.
- [Background] Kjaer P, Korsholm L, Bendix T, Sorensen JS, Leboeuf-Yde C. Modic changes and their associations with clinical findings. Eur Spine J. 2006 Sep;15(9):1312-9. doi: 10.1007/s00586-006-0185-x. Epub 2006 Aug 9. PMID 16896838
- [Background] Thompson KJ, Dagher AP, Eckel TS, Clark M, Reinig JW. Modic changes on MR images as studied with provocative diskography: clinical relevance--a retrospective study of 2457 disks. Radiology. 2009 Mar;250(3):849-55. doi: 10.1148/radiol.2503080474. PMID 19244050
- [Background] Chou R, Baisden J, Carragee EJ, Resnick DK, Shaffer WO, Loeser JD. Surgery for low back pain: a review of the evidence for an American Pain Society Clinical Practice Guideline. Spine (Phila Pa 1976). 2009 May 1;34(10):1094-109. doi: 10.1097/BRS.0b013e3181a105fc. PMID 19363455
- [Background] Resnick DK, Watters WC. Lumbar disc arthroplasty: a critical review. Clin Neurosurg. 2007;54:83-7. PMID 18504901
- [Background] Freeman BJ, Mehdian R. Intradiscal electrothermal therapy, percutaneous discectomy, and nucleoplasty: what is the current evidence? Curr Pain Headache Rep. 2008 Jan;12(1):14-21. doi: 10.1007/s11916-008-0004-7. PMID 18417018
- [Background] Helm S, Hayek SM, Benyamin RM, Manchikanti L. Systematic review of the effectiveness of thermal annular procedures in treating discogenic low back pain. Pain Physician. 2009 Jan-Feb;12(1):207-32. PMID 19165305
- [Background] Nomura T, Mochida J, Okuma M, Nishimura K, Sakabe K. Nucleus pulposus allograft retards intervertebral disc degeneration. Clin Orthop Relat Res. 2001 Aug;(389):94-101. doi: 10.1097/00003086-200108000-00015. PMID 11501830
- [Background] Okuma M, Mochida J, Nishimura K, Sakabe K, Seiki K. Reinsertion of stimulated nucleus pulposus cells retards intervertebral disc degeneration: an in vitro and in vivo experimental study. J Orthop Res. 2000 Nov;18(6):988-97. doi: 10.1002/jor.1100180620. PMID 11192261
- [Background] Ganey T, Libera J, Moos V, Alasevic O, Fritsch KG, Meisel HJ, Hutton WC. Disc chondrocyte transplantation in a canine model: a treatment for degenerated or damaged intervertebral disc. Spine (Phila Pa 1976). 2003 Dec 1;28(23):2609-20. doi: 10.1097/01.BRS.0000097891.63063.78. PMID 14652478
- [Background] Gruber HE, Johnson TL, Leslie K, Ingram JA, Martin D, Hoelscher G, Banks D, Phieffer L, Coldham G, Hanley EN Jr. Autologous intervertebral disc cell implantation: a model using Psammomys obesus, the sand rat. Spine (Phila Pa 1976). 2002 Aug 1;27(15):1626-33. doi: 10.1097/00007632-200208010-00007. PMID 12163723
- [Background] Gorensek M, Jaksimovic C, Kregar-Velikonja N, Gorensek M, Knezevic M, Jeras M, Pavlovcic V, Cor A. Nucleus pulposus repair with cultured autologous elastic cartilage derived chondrocytes. Cell Mol Biol Lett. 2004;9(2):363-73. PMID 15213815
- [Background] Meisel HJ, Siodla V, Ganey T, Minkus Y, Hutton WC, Alasevic OJ. Clinical experience in cell-based therapeutics: disc chondrocyte transplantation A treatment for degenerated or damaged intervertebral disc. Biomol Eng. 2007 Feb;24(1):5-21. doi: 10.1016/j.bioeng.2006.07.002. Epub 2006 Jul 21. PMID 16963315
- [Background] Meisel HJ, Ganey T, Hutton WC, Libera J, Minkus Y, Alasevic O. Clinical experience in cell-based therapeutics: intervention and outcome. Eur Spine J. 2006 Aug;15 Suppl 3(Suppl 3):S397-405. doi: 10.1007/s00586-006-0169-x. Epub 2006 Jul 19. PMID 16850291
- [Background] Trounson A. New perspectives in human stem cell therapeutic research. BMC Med. 2009 Jun 11;7:29. doi: 10.1186/1741-7015-7-29. PMID 19519878
- [Background] Stoyanov JV, Gantenbein-Ritter B, Bertolo A, Aebli N, Baur M, Alini M, Grad S. Role of hypoxia and growth and differentiation factor-5 on differentiation of human mesenchymal stem cells towards intervertebral nucleus pulposus-like cells. Eur Cell Mater. 2011 Jun 20;21:533-47. doi: 10.22203/ecm.v021a40. PMID 21710444
- [Background] Thompson JP, Pearce RH, Schechter MT, Adams ME, Tsang IK, Bishop PB. Preliminary evaluation of a scheme for grading the gross morphology of the human intervertebral disc. Spine (Phila Pa 1976). 1990 May;15(5):411-5. doi: 10.1097/00007632-199005000-00012. PMID 2363069
- [Background] Yamamoto Y, Mochida J, Sakai D, Nakai T, Nishimura K, Kawada H, Hotta T. Upregulation of the viability of nucleus pulposus cells by bone marrow-derived stromal cells: significance of direct cell-to-cell contact in coculture system. Spine (Phila Pa 1976). 2004 Jul 15;29(14):1508-14. doi: 10.1097/01.brs.0000131416.90906.20. PMID 15247571
- [Background] Monfort J, Garcia-Giralt N, Lopez-Armada MJ, Monllau JC, Bonilla A, Benito P, Blanco FJ. Decreased metalloproteinase production as a response to mechanical pressure in human cartilage: a mechanism for homeostatic regulation. Arthritis Res Ther. 2006;8(5):R149. doi: 10.1186/ar2042. PMID 16972994
- [Background] Murphy CL, Thoms BL, Vaghjiani RJ, Lafont JE. Hypoxia. HIF-mediated articular chondrocyte function: prospects for cartilage repair. Arthritis Res Ther. 2009;11(1):213. doi: 10.1186/ar2574. Epub 2009 Feb 5. PMID 19232075
- [Background] Salem HK, Thiemermann C. Mesenchymal stromal cells: current understanding and clinical status. Stem Cells. 2010 Mar 31;28(3):585-96. doi: 10.1002/stem.269. PMID 19967788
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Watanabe A, Benneker LM, Boesch C, Watanabe T, Obata T, Anderson SE. Classification of intervertebral disk degeneration with axial T2 mapping. AJR Am J Roentgenol. 2007 Oct;189(4):936-42. doi: 10.2214/AJR.07.2142. PMID 17885068
- [Background] Maughan EF, Lewis JS. Outcome measures in chronic low back pain. Eur Spine J. 2010 Sep;19(9):1484-94. doi: 10.1007/s00586-010-1353-6. Epub 2010 Apr 17. PMID 20397032
- [Background] Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989 Dec;10(4):407-15. doi: 10.1016/0197-2456(89)90005-6. PMID 2691207
- [Background] Stratford PW, Binkley JM, Riddle DL, Guyatt GH. Sensitivity to change of the Roland-Morris Back Pain Questionnaire: part 1. Phys Ther. 1998 Nov;78(11):1186-96. doi: 10.1093/ptj/78.11.1186. PMID 9806623
- [Background] Beurskens AJHM, de Vet HCW, Koke AJA. Responsiveness of functional status in low back pain: a comparison of different instruments. Pain. 1996 Apr;65(1):71-76. doi: 10.1016/0304-3959(95)00149-2. PMID 8826492
- [Background] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Background] Rocchi MB, Sisti D, Benedetti P, Valentini M, Bellagamba S, Federici A. Critical comparison of nine different self-administered questionnaires for the evaluation of disability caused by low back pain. Eura Medicophys. 2005 Dec;41(4):275-81. PMID 16474281
- [Background] Bombardier C, Hayden J, Beaton DE. Minimal clinically important difference. Low back pain: outcome measures. J Rheumatol. 2001 Feb;28(2):431-8. PMID 11246692
- [Background] Lauridsen HH, Hartvigsen J, Manniche C, Korsholm L, Grunnet-Nilsson N. Responsiveness and minimal clinically important difference for pain and disability instruments in low back pain patients. BMC Musculoskelet Disord. 2006 Oct 25;7:82. doi: 10.1186/1471-2474-7-82. PMID 17064410
- [Background] Perry J, Haughton V, Anderson PA, Wu Y, Fine J, Mistretta C. The value of T2 relaxation times to characterize lumbar intervertebral disks: preliminary results. AJNR Am J Neuroradiol. 2006 Feb;27(2):337-42. PMID 16484406
- [Background] Recommendations of the International Conference on Harmonization. . in Fed Regist. 1997.
- [Background] Prologo JD, Pirasteh A, Tenley N, Yuan L, Corn D, Hart D, Love Z, Lazarus HM, Lee Z. Percutaneous image-guided delivery for the transplantation of mesenchymal stem cells in the setting of degenerated intervertebral discs. J Vasc Interv Radiol. 2012 Aug;23(8):1084-1088.e6. doi: 10.1016/j.jvir.2012.04.032. Epub 2012 Jun 26. PMID 22739647
- [Background] Lalu MM, McIntyre L, Pugliese C, Fergusson D, Winston BW, Marshall JC, Granton J, Stewart DJ; Canadian Critical Care Trials Group. Safety of cell therapy with mesenchymal stromal cells (SafeCell): a systematic review and meta-analysis of clinical trials. PLoS One. 2012;7(10):e47559. doi: 10.1371/journal.pone.0047559. Epub 2012 Oct 25. PMID 23133515
- [Background] Chinnadurai R, Copland IB, Garcia MA, Petersen CT, Lewis CN, Waller EK, Kirk AD, Galipeau J. Cryopreserved Mesenchymal Stromal Cells Are Susceptible to T-Cell Mediated Apoptosis Which Is Partly Rescued by IFNgamma Licensing. Stem Cells. 2016 Sep;34(9):2429-42. doi: 10.1002/stem.2415. Epub 2016 Jul 4. PMID 27299362
- [Background] Moll G, Alm JJ, Davies LC, von Bahr L, Heldring N, Stenbeck-Funke L, Hamad OA, Hinsch R, Ignatowicz L, Locke M, Lonnies H, Lambris JD, Teramura Y, Nilsson-Ekdahl K, Nilsson B, Le Blanc K. Do cryopreserved mesenchymal stromal cells display impaired immunomodulatory and therapeutic properties? Stem Cells. 2014 Sep;32(9):2430-42. doi: 10.1002/stem.1729. PMID 24805247
- [Background] Xu X, Liu Y, Cui Z, Wei Y, Zhang L. Effects of osmotic and cold shock on adherent human mesenchymal stem cells during cryopreservation. J Biotechnol. 2012 Dec 31;162(2-3):224-31. doi: 10.1016/j.jbiotec.2012.09.004. Epub 2012 Sep 16. PMID 22989486
- [Background] Chinnadurai R, Garcia MA, Sakurai Y, Lam WA, Kirk AD, Galipeau J, Copland IB. Actin cytoskeletal disruption following cryopreservation alters the biodistribution of human mesenchymal stromal cells in vivo. Stem Cell Reports. 2014 Jun 6;3(1):60-72. doi: 10.1016/j.stemcr.2014.05.003. eCollection 2014 Jul 8. PMID 25068122
- [Background] Francois M, Copland IB, Yuan S, Romieu-Mourez R, Waller EK, Galipeau J. Cryopreserved mesenchymal stromal cells display impaired immunosuppressive properties as a result of heat-shock response and impaired interferon-gamma licensing. Cytotherapy. 2012 Feb;14(2):147-52. doi: 10.3109/14653249.2011.623691. Epub 2011 Oct 27. PMID 22029655
- [Background] Julious SA, Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005 4:287-291. doi:1 0.1002/pst.185.
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Pfirrmann CW, Metzdorf A, Zanetti M, Hodler J, Boos N. Magnetic resonance classification of lumbar intervertebral disc degeneration. Spine (Phila Pa 1976). 2001 Sep 1;26(17):1873-8. doi: 10.1097/00007632-200109010-00011. PMID 11568697
- See also: Mesoblast, I. United States FDA clears Mesoblast phase 2 trial to treat degenerative disc disease. 2011; — http://www.mesoblast.com.